CLINICAL TRIAL: NCT00868569
Title: TAC vs TACE Plus folfox4 as the Treatment of Unresectalbe Liver Metastasis of Colorectal Cancer With Resection of the Primary Tumor: a Prospective, Randomized, Control Trial
Brief Title: Transhepatic Arterial Chemotherapy (TAC) Versus Transcatheter Arterial Chemoembolization (TACE) Plus Folfox4 as the Treatment of Unresectable Liver Metastasis of Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Xujianmin, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-03
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Liver Metastasis; Colorectal Cancer
Keywords: liver metastasis; colorectal cancer; oxaliplatine; transartery chemotherapy; embolision; Unresectable Liver Metastasis of Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): folfox4 chemotherapy was done within 28 days after primary surgery. Per 3 weeks, patients will receive one cycle. After 3 cycles, patients will received transhepatic arterial chemoembolision (TACE) using oxaliplatin, fudr, mmc and iodine. Then begin folfox4 again.
  Interventions: Procedure: TACE + folfox 4
- 2 (Active Comparator): folfox4 chemotherapy was done within 28 days after primary surgery. Per 3 weeks, patients will receive one cycle. After 3 cycles, patients will received transhepatic arterial chemotherapy (TAC) using oxaliplatin, fudr and mmc. Then begin folfox4 again.
  Interventions: Procedure: TAC + folfox4

INTERVENTIONS:
Procedure: TACE + folfox 4 — tace: oxaliplatin 100mg + fudr 1g + mmc 10mg + iodine 2ml
  folfox4
  Arms: 1
Procedure: TAC + folfox4 — tac: oxaliplatin 100mg + fudr 1g + mmc 10mg
  folfox4
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether TAC plus FOLFOX4 or TACE plus folfox4 are able to improve resection rate and overall survival in patients receiving primary colorectal tumor resection than given FOLFOX4 only.

DETAILED DESCRIPTION:
We administered three cycles FOLFOX4 plus TAC(oxaliplatin,FUDR and MMC) or FOLFOX4 plus TACE(oxaliplatin,FUDR,MMC and embolision) to primary colorectal tumor resected patients with unresected liver metastasis. The study endpoints were resection rate of liver metastasis, progression-free survival, overall survival as evaluated by intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* age < 75 years with histologically proven adenocarcinoma of the colon or rectum
* no severe major organ dysfunction
* WHO performance status of 0 or 1
* no prior cancer therapy
* with measurable unresectableliver metastasis
* without other metastasis

Exclusion Criteria:

* age >= 75
* severe major organ dysfunction
* WHO performance status of >1
* prior cancer therapy
* with other metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years after operation

SECONDARY OUTCOMES:
resection rate of liver metastasis progression-free survival | 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, MD, PHD, Study Director — department of general surgery, zhongshan hospital, fudan university
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China